CLINICAL TRIAL: NCT01150396
Title: Mortality and Morbidity of Infants Born With Gestational Age Less Than 28 Weeks
Brief Title: Prognosis of Extremely Premature Birth
Acronym: BabyPEP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Bergen (Other)
Collaborators: Haukeland University Hospital (Other); Helse Stavanger HF (Other Government)
Responsible Party: Principal Investigator, Trond Markestad, Professor, University of Bergen
Other Study IDs: 2010/496
Record Dates: First submitted 2010-06-23; First posted 2010-06-25 (Estimated); Last update posted 2015-06-02 (Estimated); Status verified 2015-06

CONDITIONS: Infant, Premature, Diseases; Perinatal Morbidity; Development; Problem;Growth
Keywords: extremely premature infant; outcome; follow-up
MeSH Terms: conditions — Infant, Premature, Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood and amniotic fluid from mother Placenta Blood from umbilical cord and repeated blood samples from the infant Repeated urine samples from infant repeated tracheal spirates from the infant (while intubated)
Oversight: Data Monitoring Committee: No

SUMMARY:
Pregnant women at risk of giving birth before 28 weeks' gestational age will be enrolled. Fetal circulation will be studied and blood for inflammatory parameters will be collected. If birth occurs before 28 weeks, detailed information on clinical course of the newborn until discharge from the neonatal intensive care unit will be recorded,and specimens of amniotic fluid, placenta, blood and urine will be collection for inflammatory parameters. After discharge the children will be followed according to a specific protocol until 5 years of age.

DETAILED DESCRIPTION:
The study includes a regional cohort (Western Norway) of approximately 50 extremely preterm infants born per year over a three year period. Detailed information on fetal condition (growth, circulation, infection), neonatal resuscitation and clinical course (details on ventilatory support, circulation, pulmonary function as assessed with a neonatal spirometry technique, cerebral imaging, nutrition, growth) will be recorded. Biobank samples of blood and amniotic fluid from the mother, and from placenta, blood, urine, and tracheal aspirates will be collected form the infant, primarily to examine for inflammatory parameters. After discharge, follow-up at 6, 12, 36 and 56 months will be conducted using standardized tests (Ages & Stages, INFANIB, Denver Developmental Screening test, Bayley scales, WPPSI and ABC movement tests).

ELIGIBILITY:
Inclusion Criteria:

* Born with gestational age less than 28 weeks

Exclusion Criteria:

* None

Ages: 22 Weeks to 27 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Infants born before 28 weeks' gestational age
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2010-07; Primary Completion 2017-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Health | 40 weeks
  Outcome in terms of growth, lung function, cerebral imaging (MR), cardiac and intestinal morbidity at discharge from the neonatal intensive care unit

SECONDARY OUTCOMES:
Health | 1 year
  Growth and Developmental outcome at 12 months corrected age
Health | 3 years
  Outcome in terms of growth, behavior and psychomotor development (Bayley scales)
Health | 5 years
  Growth and motor, cognitive and mental development at 5 years of age (ABC movement test, WPPSI)

CONTACTS AND LOCATIONS:
Overall Officials: Trond Markestad, MD, PhD, Principal Investigator — University of Bergen, Faculty of Medicine
Locations (2):
- Norway (2):
  - Haukeland University Hospital, Bergen
  - Stavanger University Hospital, Stavanger

REFERENCES:
- [Derived] Bentsen MH, Markestad T, Oymar K, Halvorsen T. Lung function at term in extremely preterm-born infants: a regional prospective cohort study. BMJ Open. 2017 Oct 25;7(10):e016868. doi: 10.1136/bmjopen-2017-016868. PMID 29074512